CLINICAL TRIAL: NCT03220412
Title: Exposure to Gun Violence in Movies Increases Interest in Real Guns
Brief Title: Viewing Movie Violence & Interest in Guns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Brad Bushman, Professor of Communication & Psychology, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2013B0542-3
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Results first posted 2019-05-10 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Psychology, Social; Adolescent Behavior
Keywords: adolescent; gun; violence; media
MeSH Terms: conditions — Adolescent Behavior | interventions — Motion Pictures; Firearms

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to watch a movie containing guns, or a movie not containing guns.
Who Masked: Participant
Masking Description: Participants did not know which condition they were in. Participants' parents were aware of the deception (hidden gun) and what condition their children were in (with or without guns). Research personnel knew conditions as well. Research assistants who transcribed recorded laboratory sessions did not know what condition they were coding (eg. what type of movie participants watched)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Condition (Experimental): Intervention was guns in movies. Participants in this condition viewed a movie with guns, as it was filmed and distributed. The actual scenes in the movie (National Treasure or The Rocketeer) was not edited, but the same scenes were used as the Experimental Condition Intervention is m
  Interventions: Behavioral: Movies with Guns
- Control Condition (No Intervention): Participants in this condition viewed a movie without guns. The movie (National Treasure or The Rocketeer) was edited to remove guns from scenes.

INTERVENTIONS:
Behavioral: Movies with Guns — Participants in this arm viewed movies (National Treasure, The Rocketeer) without guns. The movies, rated PG, were edited to remove guns from the scenes
  Arms: Experimental Condition

SUMMARY:
More American children die by accidental gun use than children in other developed countries. One factor that can influence children's interest in guns is exposure to media containing guns. The objective of this study is to test whether children who see a movie containing guns will handle a real gun longer and will pull the trigger more times than children who see the same movie without guns.

DETAILED DESCRIPTION:
A recent analysis of top selling films found that the depiction of guns in violent scenes in PG-13 films that target youth has increased from the level of G and PG files in 1985 when the rating was introduced, to the level of R films by 2005, to exceed the level of R films since 2012. By definition, a PG-13 movie is supposed to have less violence than an R-rated movie. The Motion Picture Association of America says on its website that the violence in a PG-13 movie "does not reach the restricted R category." Our study shows that it does. By including guns in violent scenes, film producers may be inadvertently increasing aggression in youth via a weapons effect. This experiment directly tests this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

Age 8-12yrs, had not participated in study prior, was able to schedule participation with a known peer (8-12yo).

Exclusion Criteria:

Younger than 8yo, older than 12yo, had participated in study prior, could not schedule participation with a known peer (8-12yo)

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 104 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-01-01 (Actual); Study Completion 2016-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad J Bushman, PhD, Principal Investigator — The Ohio State Universit

IPD SHARING:
Plan to Share IPD: Undecided
We are considering making individual participant data available, but need to determine steps and appropriateness according to our institutional IRB board.

REFERENCES:
- [Derived] Dillon KP, Bushman BJ. Effects of Exposure to Gun Violence in Movies on Children's Interest in Real Guns. JAMA Pediatr. 2017 Nov 1;171(11):1057-1062. doi: 10.1001/jamapediatrics.2017.2229. PMID 28973535

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Condition: Participants in this condition viewed a movie without guns. The movie (National Treasure or The Rocketeer) was edited to remove guns from scenes.
  Movies without Guns: Participants in this arm viewed movies (National Treasure, The Rocketeer) without guns. The movies, rated PG, were edited to remove guns from the scenes
- Control Condition: Participants in this condition viewed a movie with guns, as it was filmed and distributed. The actual scenes in the movie (National Treasure or The Rocketeer) was not edited, but the same scenes were used as the Experimental Condition
Period: Overall Study
Arm/Group | Experimental Condition | Control Condition
Started | 54 | 50
Completed | 54 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Condition | Control Condition | Total
Number analyzed (Participants) | 54 | 50 | 104
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54 | 50 | 104
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (1.5) | 10.14 (1.5) | 9.9 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 26 | 42
  Male | 38 | 24 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 53 | 48 | 101
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 33 | 29 | 62
  More than one race | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 50 | 104

OUTCOME MEASURES:

1. Primary Outcome: Trigger Pulls
Description: The adjusted median of the number of trigger pulls per child. These data refer to the reduced Generalized Estimating Equation model for the two conditions. This model included participant gender and condition, bu not any of the other control variables.
Time Frame: 20 minutes after intervention
Measure: Median (95% Confidence Interval); unit: Number of trigger pulls
Groups:
- Experimental Condition: Participants in this condition watched movies as they were released, with guns.
- Control: Participants in this condition watched the same movie and same scenes with guns edited out of the scenes.
Arm/Group | Experimental Condition | Control
Number analyzed (Participants) | 54 | 50
Number of trigger pulls | 2.8 [0.2 to 2.8] | 0.01 [0.01 to 0.2]

2. Primary Outcome: Seconds Holding Gun
Description: Number of seconds participant held gun
Time Frame: 20 minutes after intervention
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Experimental Condition | Control Condition
Number analyzed (Participants) | 54 | 50
seconds | 53.1 [35.1 to 53.1] | 11.1 [10.7 to 16.7]

ADVERSE EVENTS:
Arm/Group | Experimental Condition | Control Condition
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/50
Other Adverse Events (participants affected / at risk) | 0/54 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes